CLINICAL TRIAL: NCT05526794
Title: Evaluation of Anesthesia Methods in Patients Undergoing Percutaneous Kyphoplasty: A Prospective Study
Brief Title: Anesthesia Methods on Percutaneous Kyphoplasty
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tugba Onur, Principal İnvestigator, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2021-KAEK-25 2021/12-09
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Vertebral Fracture
Keywords: percutan kyphoplasty; Vertebroplasty
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: General anesthesia or sedation
  Interventions: Procedure: Analgesic consumption
- Group 2: Central Block (Spinal and Epidural Anesthesia
  Interventions: Procedure: Analgesic consumption
- Group 3: Peripheral Block [Erector Spina Plane Block (ESPB), and Paravertebral Block (PVB)
  Interventions: Procedure: Analgesic consumption

INTERVENTIONS:
Procedure: Analgesic consumption — 1 gr iv paracetamol for all patients with a VAS value of 2 or 3; for 4 and over, 1.5 mg/kg iv tramadol was administered additionally.

SUMMARY:
The aim of this research is to examine the effects of the anesthesia method and preoperative characteristics on postoperative results and complications in patients who underwent percutaneous kyphoplasty (PKP).

Method: Patients were split into three groups according to anesthesia methods: (1) General Anesthesia (Sedation), (2) Central Block (Spinal and Epidural Anesthesia), (3) Peripheral Block [Erector Spina Plane Block (ESPB), and Paravertebral Block (PVB)]. Patients' pain values, hemodynamic parameters, additional need for sedation, and perioperative and postoperative complications were recorded prospectively together with Visual Pain Scales (VAS).

DETAILED DESCRIPTION:
Demographic characteristics (body mass index [BMI], gender, age, ASA use, pain values [VAS] before surgery, analgesic use habits, anesthesia technique chosen by anesthesiologist blind to the study, perioperative hemodynamic parameters, additional opioid during surgery, parol? or anesthetic need, perioperative complications [patients who willingly stopped the procedure during the intervention, moaning, hypotension, hypertension, bradycardia, respiratory depression, desaturation and need for mask ventilation] were taken from the records of the individuals with the treatment of PKP between 01/22-07/22 after the approval of the SBÜ Bursa Yüksek İhtisas EAH Ethics Committee (2021-KAEK-25 2021/12-09) and the patient's consent. In addition, the first mobilization time, additional analgesic need, total amount of analgesic used in 24 hours, discharge time, VAS values at 2, 6,12, and 18 hours, complications (nausea, vomiting, pain, delirium, respiratory insufficiency, infection, deep vein thrombosis, pulmonary embolus, need for re-operation, need for intensive care or mechanic ventilator) were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 ages kyphoplasty surgery patients
* written consent form received

Exclusion Criteria:

* The patient's unwillingness to participate in the study
* inability to communicate with the patient
* the patient does not speak Turkish,
* previous CVO, presence of cognitive impairment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-100 aged kyphoplasty patients
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Visual Analog Scala (VAS) values | VAS values at postoperative 24 hours
  VAS is a scala between 0-10 points. If there is no pain it means 0; very severe pain is 10 points.

SECONDARY OUTCOMES:
Analgesic consumption | postoperative 24 hours after surgery
  In all times that VAS is recorded;1 gr iv paracetamol for all patients with a VAS value of 2 or 3; for 4 and over, 1.5 mg/kg iv tramadol was administered additionally.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba T Onur, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Ümran Ü Karaca, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Asiye A Demirel, MD, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Şeyda Efsun ŞE Özgünay, Assoc Prof, Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital; Anıl A Onur, MD, Study Chair — Bursa Medicabil Hospital
Locations (1):
- Bursa Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
With the written consent of the patients and the approval of the ethics committee, I do not intend to share their special circumstances and information other than the study data.